CLINICAL TRIAL: NCT05656326
Title: Follow-up After Surgery for Colorectal Cancer: the Prospective, Multicentre FUTURE-primary Implementation Study
Brief Title: Follow-up After Surgery for Colorectal Cancer
Acronym: FUTURE-primary
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, D.J. (Dirk) Grünhagen, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL77810.078.21
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Quality of Life
Keywords: Patient-led; Home-based
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The currently developed implementation study aims to evaluate if a patient-led home-based follow-up approach is successful, improves quality of life, reduces anxiety and lessens fear of cancer recurrence during the years after surgical treatment of colorectal cancer (CRC).

DETAILED DESCRIPTION:
As the available literature implies that intensive postoperative surveillance has no impact on (cancer-specific) survival outcomes in patients after curative intent surgery for CRC, critical appraisal of the current follow-up practice and guidelines is needed. Although patients in the referenced randomized controlled trials were included roughly 5 - 15 years ago, treatment for recurrent colorectal cancer has seen little to no change since then. Therefore, efforts to improve the current standard of follow-up in patients with CRC should focus on ameliorating quality of life and cost-effectiveness, rather than survival. It provides an opportunity to support patients emotionally, to evaluate treatment effects and complications, and to inform them on their individual prognosis. This is especially true considering the growing importance of value based healthcare and patient reported outcomes in medicine. The investigators therefore propose a patient-led home-based follow-up approach. This follow-up strategy primarily consists of carcinoembryonic antigen (CEA) level monitoring at home, but additional counselling/diagnostic testing remains possible if desired by patients. In this way the investigators hope to meet the individual needs of patients during follow-up and to improve quality of life outcomes, while achieving equal or greater societal cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma without distant metastasis and treated with curative intent surgical resection less than 6 months ago
* Scheduled or currently undergoing postoperative surveillance according to national guidelines
* Written informed consent by the patient

Exclusion Criteria:

* Patients with a severely complicated postoperative course, needing in hospital follow-up longer than 6 months postoperatively
* Patients enrolled in other studies that require strict adherence to any specific follow-up practice with regular imaging - yearly or more frequent - of the abdomen and/or thorax
* Patients with comorbidity or other malignancy that requires imaging of the abdomen and/or thorax every year or more frequent
* Inability to complete the questionnaires due to illiteracy and/or insufficient proficiency of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years or older who received curative intent surgical treatment for CRC, and who (will) undergo postoperative surveillance are eligible. Patients can be included up to 6 months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Successful implementation | Year 7 (after the last follow-up moment of the last included patient)
  Patient-led follow-up will be considered successful if the used optional follow up rate is below 75%.

SECONDARY OUTCOMES:
Successful home-based sampling | Year 7
  Defined as 25% or more of all scheduled or optional CEA assessments actually performed in blood collected by the patients themselves using the self-administered blood-sampling kit
Quality of life of cancer patients | Year 7
  Measured by the EORTC Core Quality of Life questionnaire (QLQ-C30). All scales and single-item measures range from 0-100 and are calculated using their respective formulas. Higher scores mean a better outcome.
Health-related quality of life | Year 7
  Measured by the EORTC Quality of Life Questionnaire - Colorectal Cancer Module (EORTC QLQ-CR29). All scales and single-item measures range from 0-100 and are calculated using their respective formulas. Higher scores mean a better outcome.
Momentary quality of life | Year 7
  Measured by ecological momentary assessment using the Global health status of the EORTC QLQ-C30. The 2 items are scored on a Likert-scale from 1 to 7. Higher scores mean a better outcome.
Anxiety | Year 7
  Measured by The State-Trait Anxiety Inventory: Six-Item Short-form (STAI-6). The STAI-6 comprises of 6 items, each scored on a Likert-scale from 1-4. The final score ranges from 20-80 and is calculated by adding up the score of all single items (positive items are reverse scored) and multiplying by 20/6. Higher scores mean a better outcome.
Fear of cancer recurrence | Year 7
  Measured by the Assessment of Survivor Concerns - Cancer Worry subscale (ASC-CW). The total score is calculated by adding up the individual items and ranges from 3-12. Higher scores mean a worse outcome.
Cost-effectiveness of a patient-led home-based follow-up | Year 7
  The primary effect measure for the economic evaluation will be quality of life, using the The European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) as a basis for measuring utility. The EQ-5D-5L consists of five levels (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each scored on a Likert-scale from 1-5 and a visual analogue scale (VAS) scored from 0-100. The total score can be converted into an index value to be used in QALY analysis by ways of an index value calculator taking into account country-specific reference values.
Relation between coping style and follow-up preferences | Year 7
  Measured by the Threatening Medical Situations Inventory (TMSI). Total monitoring and blunting scores are obtained by summing up the relevant items, ranging from 12-60.
Satisfaction of the patient-led home-based follow-up | Year 7
  By a two-item questionnaire at the last follow-up. The first question about satisfaction consists of a scale from 1 to 10. Higher score means a better outcome. The second question is an open question whether the patient has ideas to improve the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Grünhagen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Kelly Raquel Voigt, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voigt KR, Wullaert L, Hoppener DJ, Schreinemakers JMJ, Doornebosch PG, Verseveld M, Peeters K, Verhoef C, Husson O, Grunhagen D. Patient-led home-based follow-up after surgery for colorectal cancer: the protocol of the prospective, multicentre FUTURE-primary implementation study. BMJ Open. 2023 Oct 12;13(10):e074089. doi: 10.1136/bmjopen-2023-074089. PMID 37827744
- See also: Information video FUTURE-primary — https://www.youtube.com/watch?v=ApXjUtfbNZ0